CLINICAL TRIAL: NCT05513157
Title: Investigation of Knee Hyperextension and Femoral Cartilage Thickness in Chronic Stroke Patients
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Atılım University (Other)
Responsible Party: Principal Investigator, Suleyman Korkusuz, Principal Investigator, Hacettepe University
Other Study IDs: E-59394181-604.01.02-37185
Record Dates: First submitted 2022-08-21; First posted 2022-08-24 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Stroke
Keywords: Stroke; Gait Analysis; Cartilage; Knee; Thickness; Ultrasonography
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic stroke patients with knee hyperextension: Chronic stroke patients with a maximum knee extension angle of less than 0 degrees in movement analysis
- Chronic stroke patients without knee hyperextension: Chronic stroke patients with a maximum knee extension angle greater than 0 degrees in movement analysis

SUMMARY:
It is aimed to measure knee hyperextension and knee joint cartilage thickness in chronic stroke patients and to examine the relationship between the factors affecting knee hyperextension and knee joint cartilage thickness.

This study, it is aimed to compare the knee joint cartilage thicknesses of the affected and unaffected extremities and to examine the relationship between knee hyperextension and knee joint cartilage thickness.

The second aim is to compare the knee joint cartilage thickness of the paretic and nonparetic extremities and in stroke patients with and without knee hyperextension.

The hypotheses of the study are:

Hypothesis 1;

H0: There is no difference between the knee joint cartilage thickness of the affected and unaffected extremities in chronic stroke patients with knee hyperextension.

H1: In chronic stroke patients with knee hyperextension, there is a difference between the knee joint cartilage thicknesses of the affected and unaffected extremities.

Hypothesis 2;

H0: There is no relationship between knee hyperextension during the stance phase of gait and knee joint cartilage thickness in chronic stroke patients.

H1: There is a relationship between knee hyperextension during the stance phase of gait and knee joint cartilage thickness in chronic stroke patients.

Hypothesis 3;

H0: There is no relationship between lower extremity muscle strength and spasticity and knee joint cartilage thickness in chronic stroke patients with knee hyperextension.

H1: There is a relationship between lower extremity muscle strength and spasticity and knee joint cartilage thickness in chronic stroke patients with knee hyperextension.

Hypothesis 4;

H0: There is no difference between the cartilage thickness of the knee joint in chronic stroke patients with and without knee hyperextension.

H1: There is a difference between the cartilage thickness of the knee joint in chronic stroke patients with and without knee hyperextension.

DETAILED DESCRIPTION:
Immobilization of extremities after stroke causes articular cartilage degeneration. Likewise, since patients tend to transfer weight to the non-paretic extremity, a load difference occurs between the lower extremity joints. Therefore, it is thought that the femoral cartilage thickness will be affected in stroke patients. Considering this information, it is thought that the femoral cartilage thickness will be different between the paretic and non-paretic extremities, and also between stroke patients with and without knee hyperextension in the stance phase. Accordingly, the first aim of this study is to measure knee hyperextension and femoral cartilage thickness (paretic and nonparetic side) of stroke patients. The second aim is to compare the femoral cartilage thickness of the paretic and nonparetic extremities and in stroke patients with and without knee hyperextension.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 40-65
* At least 6 months have passed since the stroke

Ambulation with or without a walking aid (walker, cane, or tripod)

* Being between 0-3 points according to the Modified Rankin Score
* Getting a score of 24 or higher on the Mini Mental Test
* Volunteering to participate in the study

Exclusion Criteria:

* Having a history of more than one stroke
* Known presence of dementia
* Having a known orthopedic, psychiatric or other neurological disease
* Having a situation that prevents communication
* Having a history of surgery involving lower extremities and gait

Ages: 40 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Stroke Patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Movement Analysis | Baseline
  Reflective signs will be placed on certain anatomical points on the participants and participants will be asked to walk at a distance of 5 meters. The three-dimensional positions of these reflective marks will be captured by the 8-camera Vicon motion capture system and recorded in the computer environment using Blade software.
Ultrasonography | Baseline
  Ultrasonographic evaluations were made by the same investigator using a linear/convex probe. In the supine position, with the knees fully flexed, the linear probe was placed axially in the suprapatellar region, and the distal femoral cartilage thickness was measured from the midpoints of the lateral femoral condyle, intercondylar area and medial femoral condyle. Outcome values were determined by taking the average of three consecutive measurements.

SECONDARY OUTCOMES:
Muscle Strength Assessment | Baseline
  Manual muscle testing will be performed on patients' lower extremity muscles (hip flexors, hip extensors, hip abductors, hip adductors, knee flexors, knee extensors, dorsiflexors, and plantar flexors). Manual muscle testing, Dr. It will be applied according to the method developed by Robert W. Lowett. According to this method, points between 0 and 5 will be given to the muscles according to the ability of the muscles to move against gravity in certain positions and the resistance of the movement against gravity.
Spasticity Assessment | Baseline
  Spasticity will be evaluated in patients' quadriceps muscle, hip extensors, hip adductors, hip internal retractors, and plantar flexors. Spasticity assessment will be made according to the Modified Ashword Scale and points will be given between 0 and 4. The method does not require any device and points are given between 0 and 4 according to the resistance of the muscles to be evaluated in the supine position against passive movement.

CONTACTS AND LOCATIONS:
Overall Officials: Kadriye Armutlu, Prof.Dr., Study Chair — Hacettepe University; Süleyman Korkusuz, MSc., Principal Investigator — Hacettepe University; Sibel Kibar, Assoc.Prof., Study Chair — Atılım University; Büşra Seçkinoğulları, MSc, Study Chair — Hacettepe University; Serdar Arıtan, Assist.Prof., Study Chair — Hacettepe University; Nihat Özgören, MSc, Study Chair — Hacettepe University; Ayla Fil Balkan, Assoc.Prof, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Altindağ, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tunc H, Oken O, Kara M, Tiftik T, Dogu B, Unlu Z, Ozcakar L. Ultrasonographic measurement of the femoral cartilage thickness in hemiparetic patients after stroke. Int J Rehabil Res. 2012 Sep;35(3):203-7. doi: 10.1097/MRR.0b013e3283532736. PMID 22555317
- [Background] Yalcin S, Kara M, Ozturk GT, Ozcakar L. Ultrasonographic measurements of the metacarpal and talar cartilage thicknesses in hemiplegic patients after stroke. Top Stroke Rehabil. 2017 Jan;24(1):1-4. doi: 10.1080/10749357.2016.1183357. Epub 2016 May 9. PMID 27159891
- [Background] Cooper A, Alghamdi GA, Alghamdi MA, Altowaijri A, Richardson S. The relationship of lower limb muscle strength and knee joint hyperextension during the stance phase of gait in hemiparetic stroke patients. Physiother Res Int. 2012 Sep;17(3):150-6. doi: 10.1002/pri.528. Epub 2011 Dec 7. PMID 22147298
- [Derived] Korkusuz S, Kibar S, Ozgoren N, Aritan S, Seckinogullari B, Balkan AF. Effect of Knee Hyperextension on Femoral Cartilage Thickness in Stroke Patients. Am J Phys Med Rehabil. 2024 May 1;103(5):371-376. doi: 10.1097/PHM.0000000000002323. PMID 37549370